CLINICAL TRIAL: NCT04622033
Title: Palmoplantar Psoriasis: Evaluating Efficacy and Clinical Photography With Brodalumab in Palmoplantar Psoriasis
Brief Title: Brodalumab in Palmoplantar Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First OC Dermatology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SILIQIISOD1
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Palmoplantar Psoriasis
MeSH Terms: interventions — brodalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Brodalumab 210mg (Experimental)
  Interventions: Biological: Brodalumab

INTERVENTIONS:
Biological: Brodalumab — brodalumab 210mg at week 0, 1, 2 and then every 2 weeks up to 24 weeks.

SUMMARY:
This is a Phase 4 single center, single-arm, open-label study that will evaluate the efficacy and safety of brodalumab in psoriasis patients as well as the impact on quality of life in addition to clinical photography. Efficacy will be evaluated by a study treatment assessor. The study includes a 30-day screening period with study visits at Week 0, 2, 4, 8, 12, 16, and 24. Study drug dosing will consist of patients self-injecting according to on-label FDA approved dosing of brodalumab 210mg at week 0, 1, 2 and then every 2 weeks thereafter for moderate to severe psoriasis patients after adequate injection training is given at study center site. Subjects will be instructed at Week 0 (pre-injection) by the site staff on how to self-inject via the dosing syringe. Study drug will be dispensed through the delineated REMS approved pharmacy. Baseline assessment will be performed at week 0 and efficacy assessments will be performed at week 4, 8, 12, 16 and 24, then every 2 weeks thereafter for palmoplantar psoriasis using approved dosing schedule for moderate to severe psoriasis. Patients will self inject after adequate injection training is given at the study center site.

ELIGIBILITY:
Inclusion Criteria:

Consent

* Subjects or their legally authorized representative must voluntarily sign and date an informed consent, approved by an independent ethics committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study-specific procedures.

Demographic and Laboratory Assessments

* Adult male or female, at least 18 years old.
* Laboratory values meeting the following criteria prior to the first dose of study drug: Serum aspartate transaminase < 3 × upper limit of normal (ULN); Serum alanine transaminase 3 2 × ULN; Serum direct bilirubin ≤ 2.0 mg/dL; except for subjects with isolated elevation of indirect bilirubin relating to a confirmed diagnosis of Gilbert syndrome; Total white blood cell count > 3,000/µL; Absolute neutrophil count > 1,500/µL; Platelet count > 100,000/µL; Hemoglobin > 8 g/dL. (Note: If an exclusionary laboratory result is obtained during the Screening period, one re-test of that particular test is allowed without repeating all other laboratory tests within the 30 day screening window. If the patient has recent laboratory examinations within 3 months, these results can be taken in lieu of screening labs. Subjects who initially do not meet all eligibility criteria for the study may be permitted to repeat the Screening Visit one time following re-consent. )
* Are willing or able to comply with procedures required in this protocol including self-administration of study drug.

Disease Activity

* Diagnosis of chronic palmoplantar psoriasis by a board certified dermatologist prior to the baseline visit.
* Subject meets the following disease activity criteria: stable palmoplantar psoriasis who are candidates for systemic or phototherapy.

Contraception

* For all females of child-bearing potential; a negative urine pregnancy test at the Screening Visit and a negative urine pregnancy test at baseline and following visits (as outlined in the Study Activity Table of this protocol) prior to the first dose of study drug.
* Female subjects must be postmenopausal OR permanently surgically sterile OR for a woman of child bearing potential be practicing at least one protocol-specified method of birth control that is effective from the baseline visit through at least 70 days (10 weeks) after the last dose of study drug
* Female who is not pregnant, breastfeeding, or considering becoming pregnant during the study or for approximately 70 days (10 weeks) after the last dose of study drug.

Contraception Recommendations:

* Contraception Requirements for Females Subjects must follow the following contraceptive guidelines as specified: Females, Non-Childbearing Potential Females do not need to use birth control during or following study drug treatment if considered of non-childbearing potential due to meeting any of the following criteria:

  * Postmenopausal, age > 55 years with no menses for 12 or more months without an alternative medical cause
  * Postmenopausal, age ≤ 55 years with no menses for 12 or more months without an alternative medical cause AND a follicule-stimulating hormone (FSH) level > 40 IU/L
  * Permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy)
  * Females who have not experienced menarche (at least one menstrual period)
* Females of Childbearing Potential

  * Females of childbearing potential must avoid pregnancy while taking study drug(s) and for at least 70 days after the last dose of study drug. Females must commit to one of the following methods of birth control:
  * Combined (estrogen and progestogen containing) hormonal birth control (oral, intravaginal, transdermal, injectable) associated with inhibition of ovulation initiated at least 1 month prior to study Baseline (Study Day 1)
  * Progestogen-only hormonal birth control (oral, injectable, implantable) associated with inhibition of ovulation initiated at least 1 month prior to study Baseline (Study Day 1)
  * Bilateral tubal occlusion/ligation (can be via hysteroscopy, provided a hysterosalpingogram confirms success of the procedure)
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Vasectomized sexual partner(s) (the vasectomized partner[s] has received medical assessment of the surgical success and is the sole sexual partner of the study subject).
  * True abstinence: Refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject.
  * Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable.
  * If required per local guidelines, male or female condom with or without spermicides OR cap, diaphragm or sponge with spermicides should be used in addition to one of the birth control methods listed above (excluding true abstinence). Contraception recommendations related to use of concomitant therapies prescribed per standard of care should be based on the local label.

Exclusion Criteria:

- Subject History

* No history of: Erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis; Active skin disease other than psoriasis that could interfere with the assessment of psoriasis; Chronic infections including human immunodeficiency virus, viral hepatitis (hepatitis B, hepatitis C), and/ or active TB. Subjects with a positive QuantiFERON®-TB /purified protein derivative (tuberculin) test result may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the subject has no evidence of active TB. If presence of latent TB is established, subjects are not required to be treated with prophylactic anti-TB therapy prior to or during the study, if the subject is considered low risk for reactivation per investigator judgment. Active systemic infection during the last 2 weeks prior to baseline visit (exception: common cold), as assessed by the investigator.
* No history of any documented active or suspected malignancy or history of any malignancy within the last 5 years except for successfully treated non-melanoma skin cancer or localized carcinoma in situ of the cervix.
* No history of clinically significant (per investigator's judgment) drug or alcohol abuse within the last 6 months.
* No history of underlying medical diseases or problems including but not limited to the following: Subject has been a previous recipient of a solid organ transplant; Evidence of a current or previous disease, medical condition (including chronic alcohol or drug abuse) other than psoriasis, surgical procedure (i.e., organ transplant), medical examination finding (including vital signs and electrocardiogram), or laboratory value at the screening visit outside the given range that, in the opinion of the investigator, is clinically significant and would make the study participant unreliable to adhere to the protocol or to complete the trial, compromise the safety of the patient, or compromise the quality of the data
* No history of an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients) and/or other products in the same class.
* No major surgery performed within 8 weeks prior to randomization or planned to be performed during the conduct of the trial (e.g., hip replacement, aneurysm removal, stomach ligation) as assessed by the Investigator.

Concomitant Medications

* No previous exposure to brodalumab.
* No use of any restricted medication as specified in the prohibited medications/therapy section or any drug considered likely to interfere with the safe conduct of the study.
* Subject must not have been treated with any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study.

Prohibited Medications and Therapy

* Prohibited medications and therapy are defined as using the following prohibited concomitant psoriasis treatments within the specified timeframe prior to Baseline Visit and throughout the study.
* Any systemic biologic to treat psoriasis: Adalimumab, infliximab or biosimilar versions within 12weeks; Etanercept or biosimilar versions within 6 weeks; Ixekizumab, secukinumab, or other IL-17 inhibitors within 16 weeks; Ustekinumab, efalizumab, guselkumab, tildrakizumab, mirikizumab, risankizumab or other IL-23 inhibitors within 24 weeks.
* Systemic non-biologic therapy for psoriasis, including but not limited to cyclosporine, corticosteroids, methotrexate, oral retinoids, apremilast, and fumaric acid derivatives within 4 weeks.
* Phototherapy treatment, laser therapy, tanning booth, or extended sun exposure that could affect disease severity or interfere with disease assessments within 4 weeks.
* Topical psoriasis treatments, including but not limited to corticosteroids, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, urea, alpha-or beta-hydroxyl acids, and medicated shampoos (for example those that contain > 3% salicylic acid, corticosteroids, coal tar or vitamin D3 analogues) within 2 weeks. Exception: Subjects are allowed to use bland (containing no psoriasis treatment) emollients and shampoos and/or low potency topical corticosteroids (US Class 6 -7) on the palms, soles, face, infra-mammary area, and groin only.
* Treatment with an experimental non-biologic for psoriasis within 4 weeks or five half-lives of the drug (whichever is longer).
* Treatment with an experimental biologic for psoriasis within 12 weeks or five half-lives of the drug (whichever is longer).
* Receipt of any live vaccine within 6 weeks or is expected to need live vaccination during study participation, including at least 20 weeks after the last dose of study drug.
* Live or attenuated vaccines are NOT allowed during the study and for 70 days after the last dose of study drug. Examples of such vaccines include but are not limited to the following: Live attenuated influenza, Herpes zoster (i.e., Zostavax®), Rotavirus, Varicella (chicken pox), Measles-mumps-rubella (MMR) or measles mumps rubella varicella (MMRV), Oral polio vaccine (OPV), Smallpox, Yellow fever, Bacille Calmette-Guérin (BCG), Oral typhoid.
* Vaccines that are inactivated, toxoid, or biosynthetic may be administered at any time without restrictions. Examples of common vaccines that meet these criteria include but are not limited to: injectable influenza vaccine, pneumococcal, pertussis (Tdap), and Shingrix®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in PASI from baseline to week 24 and the endpoint of subjects achieving palmoplantarIGA of clear (0) or almost clear (1). Lower scores are better. | 24 weeks
  Mean change in PASI from baseline to week 24 and the endpoint of subjects achieving palmoplantarIGA of clear (0) or almost clear (1). Lower scores are better.

IPD SHARING:
Plan to Share IPD: No